CLINICAL TRIAL: NCT06253013
Title: A Program of Care in Chronic Obstructive Pulmonary Disease Involving Virtual Pulmonary Rehabilitation, Integrated Care and Remote Clinical Monitoring After Discharge From a Recent Exacerbation: Mixed-Methods Study on Feasibility
Brief Title: CHARM-COPD Program of Care
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Health Network, Toronto (Other)
Collaborators: The Salvation Army Toronto Grace Health Centre (Unknown); University of Toronto (Other)
Responsible Party: Principal Investigator, Robert Wu, Doctor, University Health Network, Toronto
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 23-5062
Record Dates: First submitted 2024-01-31; First posted 2024-02-12 (Actual); Last update posted 2025-01-27 (Actual); Status verified 2025-01

CONDITIONS: Chronic Obstructive Pulmonary Disease
Keywords: Remote Clinical Monitoring; COPD; Wearables; Digital Health; Self-management
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — Sound Recordings

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Full study intervention (Experimental): In addition to the standard of care at the institutions which includes virtual pulmonary rehabilitation, remote clinical monitoring and integrated care, patients will have the option to use the following interventions:
  * FitBit wearable device with continuous monitoring for oxygen saturation and respiratory rate for 90 days
  * Hyfe cough monitoring smartwatch with continuous monitoring for 90 days
  * Home spirometer used once daily for 90 days
  * Audio recordings on a tablet once daily for 90 days
  Interventions: Device: Hyfe Smartwatch; Device: FitBit Versa 2; Device: Home Spirometer; Behavioral: Audio recording

INTERVENTIONS:
Device: Hyfe Smartwatch — Passive recording of audio with detection of explosive sounds. When explosive sounds are detected, a 0.5-1 seconds audio clip is recorded, and run through an algorithm to determine whether or not it is a cough.
Device: FitBit Versa 2 — Commercial watch with the capability to monitor vital signs including oxygen saturation, respiratory rate and heart rate. Patients will be able to view their data in the FitBit app.
Device: Home Spirometer — Patients will be able to perform spirometry testing at home. They will be able to view their data, and it will be uploaded to a dashboard for clinicians.
Behavioral: Audio recording — Patients will be asked to record several sentences which will be analyzed to detect speech patterns that may indicate changes in respiratory conditions.

SUMMARY:
The investigators' goal for this project is to evaluate the feasibility, acceptability, and actual usage of a program of care for patients with COPD recently discharged after an acute exacerbation. The program of care includes virtual pulmonary rehabilitation, integrated care, and remote clinical monitoring.

DETAILED DESCRIPTION:
The investigators' goal for this project is to evaluate the feasibility, acceptability, and actual usage of a multimodal, individualized program of care for patients with COPD recently discharged from hospital with an acute exacerbation. The program will combine elements of existing standards of care at two institutions, Toronto Grace Health Centre and University Health Network, with emerging technologies.

The investigators want to determine whether the program is considered appropriate and useful to both patients and health care providers, and whether it is feasible to implement. The investigators also want to determine whether it is feasible to conduct a large-scale randomized control trial of the program. The investigators will also explore whether each intervention reduces re-admissions to hospital.

ELIGIBILITY:
Inclusion Criteria:

* Referred to either Virtual Pulmonary Rehabilitation or Remote Clinical Monitoring at Toronto Grace Health Centre after discharge from UHN hospital with an AECOPD as defined by the clinical team

Exclusion Criteria:

* Pulmonary condition other than COPD as the main respiratory disease such as bronchiectasis or asthma
* Projected life expectancy ≤ 2 months , as determined by the clinical team
* Significant cognitive impairment and absence/inability of a family caregiver to consent and to follow study processes

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2023-09-15 (Actual); Primary Completion 2025-06 (Estimated); Study Completion 2025-06 (Estimated)

PRIMARY OUTCOMES:
Feasibility of the program and research study | 90 days
  Feasibility of the study and the program of care as determined by study participation and completion. The primary endpoints will be enrollments per month (at least 3 per study site) and data and follow up completeness (at least 75%).
Acceptability by patients and clinicians | 90 days
  Acceptability of the program as determined by patient questionnaire as well as patient and health care provider interview
Actual usage over 90 days | 90 days
  Actual usage of all program components determined objectively through logs

SECONDARY OUTCOMES:
Readmissions within 30 days | 30 days
  Readmissions to hospital within 30 days of discharge compared to control groups in past studies

CONTACTS AND LOCATIONS:
Overall Officials: Robert Wu, MD, Principal Investigator — University Health Network, Toronto
Locations (1):
- University Health Network, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: Yes
The UHN research team (principal investigator, research coordinator and other delegated research staff) will have access to all source data and documents.
  A dataset will be created with de-identified data from RCM. We will seek broad consent from participants for the future unspecified use of this data. This is in line with TCPS2 and CIHR funding guidelines to ensure data generated from this study is available to other researchers both in Canada and outside to inform improve patient, population and systems outcomes.
  The TGHC and UHN clinical teams will have access to PHI to conduct VPR and Integrated Care, and for clinical escalation when required from RCM.
  The UHN, TGHC, and U of T research teams will have access to anonymized data for analysis purposes.
Supporting Information: Study Protocol
Time Frame: Data will become available after study completion and for up to 5 years.
Access Criteria: Data will be stored and analyzed on the secure UHN server. De-identified data will be analyzed by trained study personnel at the University of Toronto.